CLINICAL TRIAL: NCT02369224
Title: Multicenter Validation of The Evergreen Myometric Strength Test for Lower Extremities (EMST-LE) in Multiple Sclerosis: Protocol for Strength Testing and Reliability Characteristics
Acronym: EMST-LE
Status: Completed | Type: Observational
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: TRB2014A
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
A Cross- Sectional study; To assess the intra-rater and inter-rater reliability of a hand-held dynamometer (HHD) in the assessment of lower extremity strength in patients with multiple sclerosis

DETAILED DESCRIPTION:
Patients will be tested at two visits separated by 1-21 days. At each visit, the patients would undergo bilateral lower extremity strength assessment by two physical therapists, independently and in the same order. Testing would include: hip flexion, knee extension, knee flexion, ankle dorsiflexion Testing performed with 1) HHD (three trials recording maximum voluntary force) and 2) manual muscle testing (MMT), British Medical Research Council grade 0-5)

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with clinically definite MS, aged ≥18, EDSS of 0-7.5
* Clinical stability defined as no MS exacerbation or change in disease modifying therapy for 30 days prior to screening.
* EDSS as described above

Exclusion Criteria:

Contraindications to Strength testing:

* Inflammatory myopathy
* Endocarditis, pericarditis or other unstable heart disease
* Cardiac surgery or myocardial infarction in the last 3 months
* Decompensated congestive heart failure
* Severe aortic stenosis
* Severe pulmonary hypertension
* Pulmonary embolus or infarction in the last 6 months
* Uncontrolled hypertension by history or by screening or baseline diastolic blood pressure >170, or systolic blood pressure > 105)
* Marfan's syndrome
* Pacemaker or cardiac defibrillator
* Concomitant neurodegenerative neurological disease, such as ALS or Parkinson Disease or hemiplegic stroke
* Females who are pregnant
* Cognitive deficits that would interfere with the subject's ability to give informed consent or perform study testing.
* Anticipated treatment with Novantrone (mitoxantrone) or cancer chemotherapy or surgical procedure during the study period
* Painful orthopedic condition affecting the lower extremities
* Any other serious and/or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who may qualify for this study will be identified in the context of clinical care at the participating sites. They may also be contacted through approved research flyers. Eligible patients may receive a copy of the informed consent form at the time of their clinic visit. Recruitment will also occur through local promotional opportunities (doctor's programs, patient education programs).
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the intra-rater and inter-rater reliability of a hand-held dynamometer (HHD) in the assessment of lower extremity strength in patients with multiple sclerosis | Patients will be tested at two visits separated by 1-21 days
  Inter-rater reliability intraclass correlation coefficient (ICC) combined for all observers (two observations per subject) for lower extremity Strength Sum Score (SSS)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, Principal Investigator — MS Center at Evergreen
Locations (1):
- MS Center at Evergreen Health, Kirkland, Washington, United States